CLINICAL TRIAL: NCT04350489
Title: Increased Levels of Interleukin-32 Isoforms Alpha, Beta, Gamma, and Delta in the Gingival Crevicular Fluid and Plasma of the Patients With Periodontitis
Brief Title: IL-32 Isoforms Levels in GCF and Plasma of the Patients With Periodontitis
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Figen Öngöz Dede, Principal Investigator, Ordu University
Other Study IDs: AP-1720
Record Dates: First submitted 2020-04-11; First posted 2020-04-17 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Periodontally healthy group
- Periodontitis: Patients with periodontitis
  Interventions: Other: Non-surgical periodontal treatment

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Conventional non-surgical periodontal treatment were performed
  Groups: Periodontitis

SUMMARY:
Interleukin (IL)-32, which has been recently reported to be associated with periodontitis, has been suggested to have pleiotropic effect due to its 9 different isoforms. The aim of this study was to investigate the levels of IL-32α, IL-32β, IL-32γ, IL-32δ isoforms in gingival crevicular fluid (GCF) and plasma before and after nonsurgical periodontal treatment in patients with periodontitis (P).Twenty-seven P and 27 periodontally healthy controls (C) were recruited in this study. Periodontitis patients were performed nonsurgical periodontal treatment. GCF and plasma sampling and clinical periodontal parameters were evaluated before and 1 month after treatment. Enzyme-linked immunosorbent assay was used to analyze the levels of IL-32α, IL-32β, IL-32γ, IL-32δ isoforms in GCF and plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 20 natural teeth, excluding third molars.
* Periodontitis patients had at least two non-adjacent sites per quadrant with probing depth (PD) ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm with gingival inflammation, and alveolar bone loss affecting >30% of the teeth, as detected on clinical and radiographical examinations.
* Periodontally healthy control group had no sign of gingival inflammation, no PD > 3mm and no evidence of attachment or bone loss

Exclusion Criteria:

* History of systemic disease.
* Regular use of any drugs which can effect the immune system or inflammatory response in the 6 months preceding the start of the study.
* Periodontal treatment during last 6 months that could affect periodontal status.
* Smoking.
* History of radiotherapy or chemotherapy.
* Current pregnancy, lactation or menopause.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. group (Control): Periodontally and systemically healthy
  2. group: Systemically healthy and periodontitis
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
IL-32 isoforms levels | baseline
  the levels of IL-32α, IL-32β, IL-32γ, IL-32δ isoforms in gingival crevicular fluid (GCF) and plasma
IL-32 isoforms levels | 1st month after treatment
  the levels of IL-32α, IL-32β, IL-32γ, IL-32δ isoforms in gingival crevicular fluid (GCF) and plasma

SECONDARY OUTCOMES:
correlation | baseline and 1st month after treatment
  the levels of IL-32α, IL-32β, IL-32γ, IL-32δ isoforms in gingival crevicular fluid (GCF) and plasma and clinical parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)